CLINICAL TRIAL: NCT03596385
Title: TREatment With Beta-blockers After myOcardial Infarction withOut Reduced Ejection fracTion
Brief Title: TREatment With Beta-blockers After myOcardial Infarction withOut Reduced Ejection fracTion"
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Centro Nacional de Investigaciones Cardiovasculares Carlos III (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REBOOT-CNIC
Record Dates: First submitted 2018-06-15; First posted 2018-07-23 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Adrenergic beta-Antagonists; Atenolol; Bisoprolol; Carvedilol; Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Beta-blocker therapy (Experimental): This is a strategy (pragmatic) trial. In patients allocated to "Beta-blocker therapy", beta blocker agent and dose are decided by treating physician.
  betablocker therapy chosen might be any of the following: atenolol bisoprolol carvedilol metoprolol nebivolol
  Interventions: Drug: Beta blocker
- Control (no beta-blocker therapy). (No Intervention): Do not receive beta -blocker therapy

INTERVENTIONS:
Drug: Beta blocker — long-term maintenance beta-blocker therapy
  Other Names: atenolol, bisoprolol, carvedilol, metoprolol, nevibolol.
  Arms: Beta-blocker therapy

SUMMARY:
REBOOT clinical trial will study whether long-term maintenance beta-blockers therapy results in a clinical benefit after heart attack without reduced left ventricular function. Half of the participants will be randomized to receive long-term beta-blocker therapy and the other half to no beta-blocker therapy after hospital discharge. All patients will be followed up for up to 5 years to determine the occurrence of adverse events (all cause mortality, re-infarction, and heart failure admission).

DETAILED DESCRIPTION:
Pragmatic, controlled, prospective, randomized, open-label, blinded endpoint clinical trial testing the benefits of beta-blocker maintenance therapy in patients discharged after an acute myocardial infarction (MI). Patients being discharged after an acute MI, with or without ST-segment elevation, and with a left ventricular ejection fraction >40%, and without history of heart failure (HF) prior to study inclusion, will be recruited. At discharge, patients will be randomized (1:1) to receive beta-blocker therapy (agent and dose according to treating physician) or no beta-blocker therapy. Primary outcome is the 5 years incidence of MACE (all cause mortality, reinfarction, heart failure admission).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Admitted for STEMI or NSTEMI and invasive management (i.e. coronary angiography during index hospitalization).
* LVEF>40% as evaluated by any imaging technique anytime during hospitalization.
* Signed informed consent

Exclusion Criteria:

* Known allergy or intolerance to beta-blockers
* Absolute contraindication to beta-blocker therapy according to treating physician judge
* Prior history of HF, Killip class on admission or during hospitalization ≥ II
* Severe valvular heart disease (> 3+ for aortic or mitral insufficiency, aortic or mitral valve area ≤1.0 cm2).
* Any condition (appart from AMI) that requires beta-blocker prescription on discharge according to treating physician judge
* Any medical condition that, in the investigator´s judgment, would seriously limit life expectancy (less than one year),
* Patients participating in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8505 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence rate of the composite of "all-cause death, nonfatal reinfarction, or heart failure hospitalization" (MACE) | 12-54 months since the beginning (median follow up anticipated 3.75 years)
  absolute number of patients experiencing deaths will be added to number of patients experiencing a non fatal reinfarction and to number of patients experiencing heart failure hospitalization.
  If a patient experience more than one of these events, only first event will be added for the sum of events
  EXAMPLE events in arm 1: 150 deaths+150 reinfarctions+150 heart failure hospitalizations= TOTAL 450 MACE (450 events/4234 patients enroled: event rate 10.63%)

SECONDARY OUTCOMES:
2.1 Incidence rate of individual components of the primary outcome. 2.2 Incidence rate of cardiac mortality. 2.3 Incidence of sustained ventricular tachycardia/ventricular fibrillation (VT/VF) and resuscitated cardiac arrest. | 12-54 months since the beginning (median follow up anticipated 3.75 years)
  Absolute number of events (% from total patients recruited) of the components of the MACE (eg number of all cause deaths (% from patients included) in active arm vs control).
  First event of each individual component counts for secondary outcome.
  EXAMPLE all cause death events in in arm 1: 200 deaths (200 events/4234 patients enroled: event rate 4.72%).
  nonfatal reinfarctions in in arm 1: 150 reinfarctions (150 events/4234 patients enroled: event rate 3.54%).
  note that in the example of the primary outcome, only 150 deaths are counted and for the secondary outcome 200. This is because in this hypothetical case, 50 deaths occurred in patients who previously experienced a nonfatal reinfarction

OTHER OUTCOMES:
3.1 Incidence of revascularizations during follow-up 3.2 Composite of cardiac death, stroke or myocardial infarction. 3.3 Safety endpoints 3.4 Quality of life and functional status (telephone evaluation): | 12-54 months since the beginning (median follow up anticipated 3.75 years)
  3.1: Absolute number of patients undergoing a revascularization procedure during follow-up (% from total patients recruited) note: revascularizations that were scheduled at patients' discharge inclusion WILL NOT be considered an event 3.2: absolute number of patients experiencing cardiac death will be added to number of patients experiencing a stroke and to number of patient experiencing a non fatal reinfarction.
  If a patient experience more than one of these events, only first event will be added for the sum of events
  3.3 3.3.1: Incidence of admission for symptomatic advanced atrioventricular (AV) block (Mobitz II or third degree). Absolute number of patients admitted for symptomatic AV block (% from total patients recruited) 3.3.2: Incidence of hospital admission for stroke: Absolute number of patients admitted for a stroke during follow-up (% from total patients recruited)
  3.4 EQ-5D questionnaire (0-100, 100 best) IIEF-5 quest (5-25, 25 best) PHQ-2 questionnaire (0-6, 6 worst)

CONTACTS AND LOCATIONS:
Overall Officials: Borja Ibañez, MD PhD FESC, Principal Investigator — CNIC
Locations (111):
- Italy (36):
  - Teresa Masselli Mascia, San Severo, Foggia
  - Ospedale Civile Santi Antonio e Biagio, Alessandria
  - Azienda Ospedaliero Universitaria Ospedali Riuniti, Ancona
  - Ospedale Civile, Baggiovara
  - Istituto Maugeri IRCCS, Bari
  - Ospedale San Paolo, Bari
  - Ospedale Maggiore, Bologna
  - A.O. Sant'Anna e San Sebastiano di Caserta, Caserta
  - Santa Margherita, Cortona
  - Ospedale di Cremona, Cremona
  - Ospedale di Desio, Desio
  - Ospedale San Giuseppe, Empoli
  - Ospedale di Vaio, Fidenza
  - Azienda Ospedaliera Universitaria - Ospedali Riuniti Foggia, Foggia
  - Ospedale C.G.Morgagni, Forlì
  - Ospedale Misericordia, Grosseto
  - Ospedale Gualdo Tadino, Gubbio
  - Ospedale Civile di Legnano, Legnano
  - Ospedale di Vizzolo Predabissi, Melegnano
  - Mario Negri, Milan
  - Ospedale San Paolo, Milan
  - Ospedale Sacro Cuore Don Calabria, Negrar
  - Ospedale San Luigi Gonzaga, Orbassano
  - Policlinico San Marco, Osio Sotto
  - Villa Sofía, Palermo, Palermo
  - P.O. di Passirana, Passirana
  - Ospedale G. da Saliceto ,Piacenza, Piacenza
  - Ospedalel Santa Maria delle Croci, Ravenna
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale Infermi di Rimini, Rimini
  - San Filippo Neri, Roma
  - Presidio Ospedaliero di Saronno, Saronno
  - Ospedale Veris Delli Ponti, Scorrano
  - Ospedale Bolognini, Seriate
  - Ospedale di Treviglio, Treviglio
  - Ospedale di Udine, Udine
- Spain (75):
  - Fundación Jiménez Díaz University Hospital, Madrid, Madrid
  - Complejo hospitalario universitario a Coruña, A Coruña
  - Txagorritxu, Alava
  - Fundacion Alcorcon, Alcorcón
  - Virgen de los Lirios de Alcoy, Alcoy
  - H. San Juan, Alicante
  - Hospital Alto del Gualdalquivir, Andújar
  - San Agustin, Avilés
  - Centro Medico Teknon, Barcelona
  - Clinic, Barcelona
  - Consorci Sanitari Integral, Barcelona
  - Germans Trias i Pujol, Barcelona
  - H. Vall d´Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital Universitario de Burgos, Burgos
  - H. Santa Lucía, Cartagena
  - Hosptial Universitario Reina Sofia, Córdoba
  - Hospital de Denia, Denia
  - Hospital universitario de Elche, Elche
  - Hospital Universitario de Vinalopo, Elche
  - H.Universitario de Elda, Elda
  - Hospital Arquitecto Macide, Ferrol
  - Hospital Galdakao Usansolo, Galdakao
  - Cabueñes, Gijón
  - Hospital San Cecilio, Granada
  - Hospital Virgen de las Nieves, Granada
  - H.U Juan Ramón Jimenez, Huelva
  - Complejo Hospitalario Universitario de Jaen, Jaén
  - Complejo Hospitalario Universitario Insular Materno Infantil, Las Palmas de Gran Canaria
  - Hospital de Leon, León
  - Hospital Universitario de Arnau de Vilanova, Lleida
  - Lucus Augusti, Lugo
  - Clinica La Luz, Madrid
  - CNIC, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Clinico, Madrid
  - Hospital Gregorio Marañon, Madrid
  - Hospital Quirón Pozuelo, Madrid
  - Ruber Internacional, Madrid
  - Ruber Juan Bravo, Madrid
  - Hospital de Manresa, Manresa
  - Hospital regional Universitario de Malaga, Málaga
  - Hospital Alvarez Buylla, Mieres
  - Rey Juan Carlos, Móstoles
  - Hospital Clinico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Central Asturias, Oviedo
  - Son Espases, Palma de Mallorca
  - Complejo Hospitalario de Navarra, Pamplona
  - Montecelo, Pontevedra
  - Clinico Universitario de Salamanca, Salamanca
  - Complejo hospitalario Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital General de La Palma, Santa Cruz de Tenerife
  - Nuestra Señora de la Candelaria, Santa Cruz de Tenerife
  - Marques de Valdecilla, Santander
  - Complejo hospitalario universitario de Santiago, Santiago de Compostela
  - H. Virgen del Rocio, Seville
  - Virgen de la Macarena, Seville
  - Hospital Universitari Joan XXIII, Tarragona
  - Hospital Universitario Sant Joan de Reus, Tarragona
  - Hospital Universitario de Torrejon, Torrejón de Ardoz
  - Hospital Universitario de Torrevieja, Torrevieja
  - H. Verge de la Cinta, Tortosa
  - San Juan de la Cruz, Úbeda
  - Hospital Infanta Elena, Valdemoro
  - Hospital Clinico, Valencia
  - Hospital La Fe, Valencia
  - Hospital universitario doctor Peset, Valencia
  - IMED Valencia, Valencia
  - Hospital Clinico universitario de Valladolid, Valladolid
  - Río Hortega, Valladolid
  - Alvaro Cunqueiro, Vigo
  - Hospital General de Villalba, Villalba
  - Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossello X, Raposeiras-Roubin S, Latini R, Dominguez-Rodriguez A, Barrabes JA, Sanchez PL, Anguita M, Fernandez-Vazquez F, Pascual-Figal D, De la Torre Hernandez JM, Ferraro S, Vetrano A, Perez-Rivera JA, Prada-Delgado O, Escalera N, Staszewsky L, Pizarro G, Aguero J, Pocock S, Ottani F, Fuster V, Ibanez B; REBOOT-CNIC investigators. Rationale and design of the pragmatic clinical trial tREatment with Beta-blockers after myOcardial infarction withOut reduced ejection fracTion (REBOOT). Eur Heart J Cardiovasc Pharmacother. 2022 May 5;8(3):291-301. doi: 10.1093/ehjcvp/pvab060. PMID 34351426
- [Derived] Ibanez B, Latini R, Rossello X, Dominguez-Rodriguez A, Fernandez-Vazquez F, Pelizzoni V, Sanchez PL, Anguita M, Barrabes JA, Raposeiras-Roubin S, Pocock S, Escalera N, Staszewsky L, Perez-Garcia CN, Diez-Villanueva P, Perez-Rivera JA, Prada-Delgado O, Owen R, Pizarro G, Caldes O, Gomez-Talavera S, Tunon J, Bianco M, Zarauza J, Vetrano A, Campos A, Martinez-Huertas S, Bueno H, Puentes M, Grigis G, Bonilla-Palomas JL, Marco E, Gonzalez-Juanatey JR, Bangueses R, Gonzalez-Juanatey C, Garcia-Alvarez A, Ruiz-Garcia J, Carrasquer A, Garcia-Rubira JC, Pascual-Figal D, Tomas-Querol C, San Roman JA, Baratta P, Aguero J, Martin-Reyes R, Colivicchi F, Ortas-Nadal R, Bazal P, Cordero A, Fernandez-Ortiz A, Basso P, Gonzalez E, Poletti F, Bugani G, Debiasio M, Cosmi D, Navazio A, Bermejo J, Tortorella G, Marini M, Botas J, de la Torre-Hernandez JM, Ottani F, Fuster V; REBOOT-CNIC Investigators. Beta-Blockers after Myocardial Infarction without Reduced Ejection Fraction. N Engl J Med. 2025 Nov 13;393(19):1889-1900. doi: 10.1056/NEJMoa2504735. Epub 2025 Aug 30. PMID 40888702
- [Derived] Granger CB, Pocock SJ, Gersh BJ. The need for new clinical trials of old cardiovascular drugs. Nat Rev Cardiol. 2023 Feb;20(2):71-72. doi: 10.1038/s41569-022-00819-1. No abstract available. PMID 36526898